CLINICAL TRIAL: NCT00028548
Title: Phase I Study of R(+)-XK469 (NSC 698215) Given Daily, Days 1-5, Repeated Every Three Weeks in Patients With Advanced Malignancies
Brief Title: XK469 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patricia LoRusso, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069103; U01CA062487 (NIH); P30CA022453 (NIH); WSU-C-2346; NCI-4550; WSU-T-2001
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — XK 469

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XK469 (Experimental)
  Interventions: Drug: R(+)XK469

INTERVENTIONS:
Drug: R(+)XK469

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of XK469 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, dose-limiting toxicity, and recommended phase II dose of XK469 in patients with advanced solid tumors.
* Determine the safety of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine, preliminarily, any anti-tumor activity of this drug in these patients.
* Determine the drug metabolism, drug interaction potential, molecular and cellular predictors of efficacy and toxicity, and clinical confirmation of molecular responses in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive XK469 IV over 20 minutes on days 1-5. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of XK469 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of the first 6 patients experience dose-limiting toxicity.

Once the MTD is determined, up to 15 patients are treated at that dose. Patients in the expanded MTD cohort also receive oral NovaSoy® soybean extract twice daily for the study duration.

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: Approximately 25-40 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-hematological cancer that is unresponsive to available therapies or for which there is no known effective treatment
* Measurable or evaluable disease

  * Clinical or radiological evidence of disease required
* No active brain metastases

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* Ejection fraction at least 50%
* No significant arrhythmias
* No congestive heart failure

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No dementia or altered mental status
* No known HIV infection
* No active infection
* No other serious uncontrolled medical disorder that would preclude study participation
* No known allergies to soy products, rice flour, or gelatin (if receiving study dietary soy supplementation)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent prophylactic colony-stimulating factors

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Prior taxanes allowed
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except hormone replacement therapy or medication used to maintain castrate status for patients with progressive hormone-refractory prostate cancer

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow-containing areas
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 4 weeks since prior investigational agents
* No other concurrent experimental anticancer therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. LoRusso, DO, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States